CLINICAL TRIAL: NCT03005951
Title: The Influence of Breakfast on Hormone Responses and Cognitive Performance, as Assessed by CTET in Lean and Obese Adolescent Males
Brief Title: The Influence of Breakfast on Hormone Responses and Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: New York State Department of Health (Other Government); Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2015-5542
Record Dates: First submitted 2016-06-24; First posted 2016-12-30 (Estimated); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lean males (Experimental): This is a randomized, two-period, cross over design with the intervention of consuming breakfast versus fasting for breakfast to study the effects on hormone responses and cognitive function using CTET in lean and obese male adolescents. These two study groups will be randomized to one of two orders:: (A,B) or (B,A) where A = Yes breakfast and B=No breakfast
  Interventions: Other: A= Yes Breakfast; Other: B=No Breakfast
- Obese males (Experimental): This is a randomized, two-period, cross over design with the intervention of consuming breakfast versus fasting for breakfast to study the effects on hormone responses and cognitive function using CTET in lean and obese male adolescents. These two study groups will be randomized to one of two orders:: (A,B) or (B,A) where A = Yes breakfast and B=No breakfast
  Interventions: Other: A= Yes Breakfast; Other: B=No Breakfast

INTERVENTIONS:
Other: A= Yes Breakfast — Study visit will include analysis of cognitive function (CTET), insulin, glucagon, C-peptide, free fatty acids, and GLP-1 when given breakfast and lunch
Other: B=No Breakfast — Study visit will include analysis of cognitive function (CTET), insulin, glucagon, C-peptide, free fatty acids, and GLP-1 when breakfast is skipped and lunch is provided.

SUMMARY:
The purpose of this study is to see what effect skipping breakfast versus consuming breakfast has on cognitive performance and the hormones responsible for glucose homeostasis in lean and obese adolescent males. The subjects will be tested on their ability to maintain attention when given several tasks called continuous temporal expectancy tasks (CTET) and electrophysiological signals using electroencephalogram (EEG) will be monitored. These two study groups will be randomized to one of two orders: (A,B) or (B,A) where A = breakfast intervention and B = no breakfast. There will be a washout period of 7 days in between study visits.

DETAILED DESCRIPTION:
Eating unhealthy foods and not exercising regularly contributes to obesity in children. Other unhealthy behaviors, such as skipping meals can also lead to obesity. Breakfast is known to be the most important meal of the day, yet many people skip breakfast. Skipping breakfast can cause an imbalance in the hormones that control blood glucose.

Skipping breakfast can affect how well insulin works at lowering blood glucose at later meal times. The impact of breakfast on glucose homeostasis is different from that of lunch and dinner. This became evident when a group of researchers studied the effect of skipping breakfast on hormone responses after subsequent isocaloric lunch and dinner in adults with Type 2 diabetes. The study showed that in Type 2 diabetics, skipping breakfast leads to increased post-prandial hyperglycemia and decreased glucagon-like peptide-1 (GLP-1) release, impairing the insulin response to hyperglycemia. Plasma free fatty acids (FFA) levels were found to be significantly higher after lunch and dinner when breakfast was omitted. It has been shown that acute elevation of FFA induces hepatic insulin resistance and increased hepatic glucose production in patients with Type 2 Diabetes Mellitus and in non-diabetic controls. Impaired insulin secretion can predispose to conditions such as obesity, and other diseases.

Skipping breakfast can also have a negative effect on children's ability to keep focus and attention. The CTET is a tool that can be used to directly measure attention using an EEG and is a highly sensitive measure of neural processing.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males
2. No history of neurological or psychiatric illness, including major depressive disorder and attention deficit disorder.
3. Normal or corrected vision using the Snellen chart
4. Normal hearing
5. BMI greater than or equal to 95th percentile according to the Center for Disease Control and Prevention (CDC) growth charts
6. HbA1C less than or equal to 5.6%
7. Hemoglobin level of greater or equal to 12g/dL

Exclusion Criteria:

1. History of chronic illness and chronic use of medications that affect cognitive or glucose metabolism
2. History of substance, nicotine or alcohol dependence as assessed by CRAFFT (CAR, RELAX, ALONE, FORGET, FRIENDS, TROUBLE) questionnaire
3. History of eating disorder as assessed by the SCOFF questionnaire.
4. Developmental delay
5. Hearing and vision problems as assessed by the Snellen chart
6. Previous history of bariatric surgery
7. Currently taking supplements or medications indicated for weight loss
8. Previous history of head injury associated with loss of consciousness for several minutes
9. History of Epilepsy
10. Allergy to any of the foods used for the test breakfasts

The inclusion and exclusion criteria for lean subjects will be identical to that of obese subjects with the exception that the lean subjects will be less than or equal to the 85th percentile for BMI, according to CDC growth charts.

Ages: 13 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
The measurement of glucose will be euglycemic during the breakfast study visit | 0min to 420 min during both during the treatment and control visits over the one year study period. Each study visit will be conducted on 2 separate days with a washout period of at least 1 week in between the study visits for each patient
  Area under the curve of glucose from time 0min to 420 min.
The measurement of C-peptide will be steady during the breakfast study visit | 0min to 420 min during both during the treatment and control visits over the one year study period. Each study visit will be conducted on 2 separate days with a washout period of at least 1 week in between the study visits for each patient
  Area under the curve of C-peptide from time 0min to 420 min.
The measurement of insulin will be steady during the breakfast study visit | 0min to 420 min during both during the treatment and control visits over the one year study period. Each study visit will be conducted on 2 separate days with a washout period of at least 1 week in between the study visits for each patient
  Area under the curve of insulin from time 0min to 420 min.
The measurement of free fatty acids will be steady during the breakfast study visit | 0min to 420 min during both during the treatment and control visits over the one year study period. Each study visit will be conducted on 2 separate days with a washout period of at least 1 week in between the study visits for each patient
  Area under the curve of free fatty acids from time 0min to 420 min.
The measurement of glucagon-like peptide will be steady during the breakfast study visit | 0min to 420 min during both during the treatment and control visits over the one year study period. Each study visit will be conducted on 2 separate days with a washout period of at least 1 week in between the study visits for each patient
  Area under the curve of glucagon- like peptide from time 0min to 420 min.
The measurement of glucagon will be steady during the breakfast study visit | 0min to 420 min during both during the treatment and control visits over the one year study period. Each study visit will be conducted on 2 separate days with a washout period of at least 1 week in between the study visits for each patient
  Area under the curve of glucagon from time 0min to 420 min.
The measurement of CTET will be better during the breakfast study visit | 0min to 420 min during both during the treatment and control visits over the one year study period. Each study visit will be conducted on 2 separate days with a washout period of at least 1 week in between the study visits for each patient
  Area under the curve of CTET from time 0min to 420 min.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Underland, MD, Principal Investigator — Albert Einstein College of Medicine Montefiore Medical Center
Locations (1):
- Montefiore Medical Center of Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jakubowicz D, Wainstein J, Ahren B, Landau Z, Bar-Dayan Y, Froy O. Fasting until noon triggers increased postprandial hyperglycemia and impaired insulin response after lunch and dinner in individuals with type 2 diabetes: a randomized clinical trial. Diabetes Care. 2015 Oct;38(10):1820-6. doi: 10.2337/dc15-0761. Epub 2015 Jul 28. PMID 26220945